CLINICAL TRIAL: NCT01439386
Title: Impact Of Different Ablation Approaches on Outcome In Coexistent Atrial Fibrillation and Flutter
Acronym: APPROVAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Collaborators: Monzino Hospital, Milan, Italy (Unknown); Ospedale dell'Angelo, Venezia-Mestre (Other); Catholic University, Italy (Other); University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Andrea Natale, Executive medical director, Texas Cardiac Arrhythmia Research Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCAI_APPROVAL
Record Dates: First submitted 2011-09-21; First posted 2011-09-23 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Atrial Arrhythmia; Quality of Life
MeSH Terms: interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AF ablation with or without AFL ablation (Active Comparator): Pulmonary vein antral isolation (PVAI)with or without cavo-tricuspid isthmus (CTI) ablation
  Interventions: Procedure: Catheter ablation
- AFL ablation only (Active Comparator): Cavo-tricuspid isthmus ablation only
  Interventions: Procedure: Catheter ablation

INTERVENTIONS:
Procedure: Catheter ablation — PVAI with or without CTI ablation
  Arms: AF ablation with or without AFL ablation
Procedure: Catheter ablation — CTI ablation only
  Arms: AFL ablation only

SUMMARY:
This prospective, multi-center, single blinded study aims to compare the influence of two different catheter ablation strategies, on long-term ablation outcome in terms of AF recurrence and quality of life (QoL) in patients presenting with coexistent AF and AFL. The two strategies to be evaluated are 1) the ablation of paroxysmal atrial fibrillation (PAF) with or without flutter (AFL) ablation (AF ± AFL) versus 2) AFL ablation alone.

DETAILED DESCRIPTION:
Specific Aim: This prospective single blinded study aims to compare the influence of two different catheter ablation strategies, on long-term ablation outcome in terms of AF recurrence and quality of life (QoL) in patients presenting with coexistent AF and AFL. The two strategies to be evaluated are 1) the ablation of paroxysmal atrial fibrillation (PAF) with or without flutter (AFL) ablation (AF ± AFL) versus 2) AFL ablation alone.

Hypothesis: Ablation of AF ± AFL results in better long-term procedure outcome than AFL-ablation alone in patients with a documented history of AF and AFL.

Background: Coexistence of AF and AFL is commonly encountered in clinical practice. Patients with these arrhythmias experience symptoms such as palpitation which is often described as a sudden irregular fluttering sensation in the chest, dyspnea, fatigue, dizziness and fainting attacks. These symptoms make the patients anxious and tired and seriously compromise their QoL (1).

Radiofrequency catheter ablation (RFCA) has emerged as the best therapeutic option in drug-refractory AF cases and often used as a first-line therapy in AFL (2). Several studies have demonstrated significant improvement in QoL following catheter ablation (CA) when patients have either AF or AFL (3-9). However, very little is known about the impact of CA on QoL in patients presenting with coexistent AF and AFL.

No standard treatment guidelines exist for coexistent AF and AFL. Determining the best ablative approach for this type of patient remains a challenge. Roithinger et al (10) postulated that the mechanism of AFL in patients presenting with both arrhythmias could be organization of AF to AFL. However, it is not always possible to determine which is the predominate arrhythmia. In some cases, AFL ablation can eliminate AF and AFL, and is a less extensive procedure than AF ablation. As the two arrhythmias are inter-twined, it is possible that AFL ablation alone may be sufficient to cure both arrhythmias. Should an AF ablation be required at a later date, there is no supportive data suggesting that the second procedure is associated with additional complications. Therefore, performing an AFL ablation alone does not expose the patient to any unwarranted risk. (11) Several published studies have reported on a variety of ablation strategies for different types of AF, to include paroxysmal, persistent and long standing persistent, with variable results on AF recurrence. (12-16) Compared to previous studies, the scope of the APPROVAL study is narrowed to include patients with AF falling into the 'paroxysmal' category.

In a randomized trial, Wazni et al compared the outcome in PV disconnection alone for AF versus PV disconnection plus cavotricuspid isthmus ablation for AFL. They concluded that in patients with coexistent AF and AFL, comparable long-term outcome in terms of arrhythmia-free existence was observed among patients undergoing either AF ablation only or AF+AFL ablation. Performance or lack of performance of AFL ablation along with AF ablation, did not significantly affect the long-term outcome. Therefore, the APPROVAL study allows group 1 patients to undergo the AFL ablation or not undergo the AFL ablation based on physician discretion, with the belief that an AFL ablation in this setting will not affect the outcome. Ablation of AFL for the treatment of AF / AFL, followed by anti-arrhythmic drug (AAD) therapy for 3 months is a commonly used approach. QoL assessment focuses on the physical, social and emotional consequences of illness. The subjective perception of 'illness intrusiveness', and how the disease burden affects the general well-being are of great interest in this population.(17) Several standardized questionnaires are available to quantitatively assess QoL. In this study, 4 of those will be used, namely Medical Outcome Study Short Form-36 (SF-36), Hospital Anxiety and Depression Score (HAD), Beck Depression Inventory (BDI) and State-Trait Anxiety Inventory (STAI).

Study Objective:

To compare long-term procedure-outcome, following AF with or without AFL ablation versus AFL ablation alone, in patients presenting with both PAF and AFL.

Study Design:

This prospective, single blind randomized study would enroll 86 patients presenting with documented symptomatic PAF and typical isthmus dependent AFL that are scheduled to undergo catheter ablation.

Endpoints:

Primary: Recurrence of atrial arrhythmia: any episode of AF/AT longer than 30 sec will be considered as a recurrence. Episodes that occur during the first 3 months after the procedure (blanking period) will not be considered as recurrence.

Secondary: Change in QoL score from baseline

Study Procedures:

Baseline:

Consenting patients would be randomly assigned to either AF±AFL ablation (group 1) or AFL ablation only (group 2). In group 1, AF ablation will be performed in all cases. In addition, the physician will also perform an AFL ablation if any one of the following criteria are met:

* The patient demonstrates spontaneous right-sided isthmus-dependent flutter upon arrival for the ablation procedure
* Right-sided isthmus-dependent flutter is inducible anytime during the ablation procedure
* The patient spontaneous converts to right-sided isthmus-dependent flutter anytime during the ablation procedure

In group 2, all patients will undergo ablation of AFL only. Because QoL could be affected by a placebo effect of the procedure, the patients will be blinded to their group assignment. Baseline QoL surveys will be collected for all patients prior to their ablation.

Ablation Procedure:

Standard mapping and ablation techniques will be conducted at the discretion of the physician, with RF lesions administered at the location determined by the randomization assignment. This includes pulmonary vein isolation (PVI) and ablation of extra-pulmonary triggers detected by standard mapping procedure for AF (18) and cavo-tricuspid isthmus ablation for atrial flutter (2). The endpoint of the procedure is defined as the termination or non-inducibility of AF or AFL.

Follow-up:

Study follow-up will last for one year. Following ablation, patients will be discharged on their previously ineffective AADs which will be continued for 90 days (blanking period). The blanking period allows time for the inflammatory process to subside. AADs will be discontinued after the blanking period for all patients. If a patient suffers a recurrence of an atrial arrhythmia, the primary end point will be met and the AAD therapy may be administered at the discretion of the physician.

Patients will use an event recorder for 5 months after ablation, and will be asked to transmit their rhythm every time they experience symptoms compatible with arrhythmias, and at least twice a week even if asymptomatic. Any episode of AF/AT longer than 30 sec after the 3 month blanking period will be considered as a recurrence.

A 7 day Holter monitor will be worn at the 3, 6, 9 and 12 month time points after the procedure.

QoL surveys will be self-administered at the 3 and 12-month time points.

Risk Analysis:

This study does not pose any additional risk to the patient. The risks are the same for both groups and are the same as those for a standard atrial fib or flutter ablation. Per standard of care, ablation procedures are not scheduled for pregnant patients. A pregnancy test is routinely performed prior to the ablation procedure to confirm that the patient is not pregnant.

There is no risk associated with study withdraw since the study is collecting only routine data, and there are no protocol specific follow-up procedures.

Probability of requiring a repeat ablation:

The probability of arrhythmia recurrence (AF and/or AFL) after AF ± AFL ablation was reported to be between 52% [Scharf et al (19)] to 58% [Husser et al (20)]. According to Scharf et al, the recurrence of typical flutter alone after AF ± AFL ablation was 12%.

The recurrence of typical flutter among patients undergoing AFL ablation alone, has been reported to be 11% [Bertaglia et al (21)] to 12% [Luca CT et al (22)]. However, the cumulative probability of recurrence of combined AF and AFL in this AFL ablation only population has been 50% at 2 years and 58% at 3 years.(21) Therefore, the overall probability of going for a redo ablation after AF ± AFL ablation compared to that of AFL ablation alone is not be significantly different (52% vs 50%, p>0.5).

Regarding risks associated with a repeat procedure, no additional identifiable risks have been reported for patients undergoing a second procedure (19) (23). However, potential study subjects will be advised that standard procedural risks would be present with a repeat procedure. These include cardiac tamponade CVA, esophageal fistula, pulmonary vein stenosis, bleeding, myocardial infarction, death and injury to the cardiac conduction system.

Benefits: The subject may not incur any benefit by participating in this study.

Statistical Methodology:

Sample size determination and power analysis:

Reported success rates from previous studies were used to determine the minimal difference of outcome (effect size). Published results indicate that the observed success rate (freedom from arrhythmia) has been 65% in group 1 and 30% in group 2. The sample size necessary to detect an effect size of 35% for the primary outcome was determined using alpha = 0.05 and power = 0.80 (beta= 0.20). The minimum required sample size (two-sample parallel design test for superiority model) for each group came out to be 43 patients.

Sampling Plan:

A central database will be created which will hold all the eligible subjects. Permuted block randomization method will be used for treatment allocation.

Analysis Plan:

The continuous variables will be reported as mean ± standard deviation (SD). The categorical variables will be reported as number of cases (n) and percentage. The bivariate analyses for comparing the characteristics across the two study groups will be performed using Student's t-test for continuous variables and chi-square test for categorical variables. A stratified sub-analysis will be performed for assessing outcome across AF and AF+CTI groups with a multivariable risk-adjusted model. A two-tailed p value of <0.05 is considered statistically significant. Time series analysis will be performed, using Kaplan Meier test and multivariate analysis with Cox proportional-hazards model, to compare recurrence at follow-up. SAS 9.2 (SAS Institute Inc., Cary, NC) will be used for statistical analysis. Statistical testing will compare Group 1 & 2, as well as provide a subanalysis of Group 1 (with and without AFL ablation).

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18years
2. Patients presenting with paroxysmal AF and typical AFL
3. Ability to provide written, informed consent

Exclusion Criteria:

1. Reversible causes of atrial arrhythmia such as hyperthyroidism, pneumonia, pulmonary embolism, sarcoidosis and excessive alcohol consumption
2. Bleeding disorder
3. Contra-indication to anti-coagulants

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Recurrence of atrial arrhythmia | 12 months
  Any episode of AF/AT longer than 30 sec will be considered as a recurrence. Episodes that occur during the first 3 months after the procedure (blanking period) will not be considered as recurrence.

SECONDARY OUTCOMES:
Change in QoL score from baseline | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation
Locations (1):
- Texas Cardiac Arrhythmia Institute, St. David's Medical Center, Austin, Texas, United States

REFERENCES:
- [Result] References: Symptomatic improvement after radiofrequency catheter ablation for typical atrial flutter; Heart 2001;86:167-171 Quality-of-Life in Patients With Paroxysmal Atrial Fibrillation After Catheter Ablation: Results of Long-Term Follow-Up; PACE 2003; 26:678-684 Quality of life restored to normal in patients with atrial fibrillation after pulmonary vein ostial Isolation; Am Heart J 2004;148:318-25 Effect of Left Atrial Ablation on the Quality of Life in Patients With Atrial Fibrillation; Circ J 2008; 72: 582-587 Catheter Ablation for Atrial Fibrillation in Congestive Heart Failure; N Engl J Med 2004;351:2373-83. Effects of Radiofrequency Catheter Ablation on Quality of Life in Patients With Atrial Flutter; Am J Cardiol 1999;84:278-283 Radiofrequency Catheter Ablation of Common Atrial Flutter : Significance of Palpitations and Quality-of-Life Evaluation in Patients With Proven Isthmus Block; Circulation 1999;99;534-540 Relationship Between Atrial Fibrillation and Typical Atrial Flutter in Humans; Circulation. 1997;96:3484-3491 Combining ablation of atrial fibrillation with ablation of atrial flutter: Are we there yet? JACC, Vol 43, No. 11, 2004 Factors predicting recurrences of atrial fibrillation after radiofrequency catheter ablation of typical atrial flutter; Seminars in Cardiology, 2003, vol. 9, No. 3: 55-60 Effectiveness of catheter ablation for coexisting atrial fibrillation and atrial flutter; Am J Cardiol 2004; 94:666-668 Quality of Life in Atrial Fibrillation: Measurement Tools and Impact of Interventions; J Cardiovasc Electrophysiol. 2008 July ; 19(7): 762-768 Clinical significance of inducible atrial flutter during pulmonary vein isolation in patients with atrial fibrillation. J Am Coll Cardiol. 2004 Jun 2;43(11):2057-62. Effectiveness of catheter ablation for coexisting atrial fibrillation and atrial flutter. Am J Cardiol. 2004 Sep 1;94(5):666-8.
- [Derived] Mohanty S, Mohanty P, Di Biase L, Bai R, Santangeli P, Casella M, Dello Russo A, Tondo C, Themistoclakis S, Raviele A, Rossillo A, Corrado A, Pelargonio G, Forleo G, Natale A. Results from a single-blind, randomized study comparing the impact of different ablation approaches on long-term procedure outcome in coexistent atrial fibrillation and flutter (APPROVAL). Circulation. 2013 May 7;127(18):1853-60. doi: 10.1161/CIRCULATIONAHA.113.001855. Epub 2013 Apr 9. PMID 23572499